# COMPARISON OF CLINICAL PERFORMANCE OF LMA PROTECTOR $^{\text{TM}}$ CUFF PILOT AND LMA SUPREME AMONG ANAESTHETISED, NON-PARALYSED PATIENTS

DR. CHAN WENG KEN
M.D. (UNIMAS)

# UNIVERSITI KEBANGSAAN MALAYSIA

14 JULY 2018

#### INTRODUCTION

The inception of supraglottic airway (SGA) has revolutionized the anaesthetist's airway armamentarium. It was invented by Dr Archie Ian Jeremy Brain in 1982 and was commercially made available in 1987.<sup>1</sup> It offers the advantage of avoiding endotracheal intubation, shorter insertion time, lower incidence of post-operative pharyngeal pain and better haemodynamic stability during induction and emergence.<sup>2</sup> An ideal SGA placement should provide sufficient perilaryngeal seal to allow ventilation of the lungs without injuring pharyngeal mucosa and able to prevent or provide early detection of gastric aspiration. It can be classified based on its function into 1<sup>st</sup>, 2<sup>nd</sup> and 3<sup>rd</sup> generation<sup>3</sup> or via its sealing mechanism.<sup>4</sup>

LMA Supreme<sup>™</sup> is a single use, second generation SGA introduced in 2005. It is made of polyvinyl chloride (PVC). It has the advantage of anatomically shaped airway tube, presence of an integral bite block and a drain tube to facilitate placement of gastric tube.<sup>5</sup> According to manufacturer, it is a high volume low pressure cuff which can generate high seal pressure up to 37 cmH<sub>2</sub>O.<sup>6</sup>

LMA Protector<sup>TM</sup> is the latest second generation SGA introduced in 2015. It is a single use device made of silicon and is both latex and phthalate free. It is similar to LMA Supreme<sup>TM</sup> that has a dynamic curve, which conforms to the anatomical contour of the pharynx, hence allowing rapid insertion. LMA Protector<sup>TM</sup> also has an integral bite block and dual gastric access. In addition, LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> has an integrated cuff pressure monitor to ensure the SGA is properly inflated.<sup>7</sup>

The common complications of SGA are malposition, sore throat, dysphagia and laryngeal nerve injury.<sup>8</sup> Instruction leaflet for LMA Supreme<sup>TM</sup> states a maximum cuff volume of 20 ml, 30 ml and 40 ml of air for size 3, 4, and 5 respectively. It also recommends maximum intra-cuff pressure of 60 cmH<sub>2</sub>O.<sup>5</sup> However, inflating the maximum recommended cuff volume often results in intra-cuff pressure higher than 60 cmH<sub>2</sub>O.<sup>9,10</sup> Saraçoğlu *et al.* reported that professional experience does not contribute to obtaining optimal cuff pressure without measuring it.<sup>11</sup> Hence, this calls for a need to introduce cuff manometer into our routine anaesthetic practice.

The new LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> was designed to reduce the risk of overinflating. It has a cuff pilot valve to allow user to monitor the intra-cuff pressure of the SGA through visual means that are colour coded. Optimal intra-cuff pressure of 40-60 cmH<sub>2</sub>O will place the cuff pilot valve in green zone whereas underinflating and overinflating will place it either in yellow or red zone respectively. As it is made of silicone, it also offers more flexibility and potentially less traumatic than LMA Supreme<sup>TM</sup>. <sup>12</sup>

A search of 'LMA Protector, laryngeal mask airway protector' in PubMed Central only yielded six results, whereas 'laryngeal mask airway supreme' yielded 160 results in PubMed and 188 results in PubMed Central respectively. Only two papers mentioned LMA Protector<sup>TM</sup>'s clinical performance whereas another three were case reports. Hence, this calls for more study on LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> especially in regards to its clinical performance.

#### **OBJECTIVES**

## **Primary objective:**

To assess the oropharyngeal leak pressure (OLP) of LMA Protector<sup>TM</sup>  $Cuff Pilot^{TM}$  and LMA Supreme<sup>TM</sup>.

#### **Secondary objectives:**

- 1. To compare the mean time to insertion between LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> and LMA Supreme<sup>TM</sup>.
- 2. To compare the ease of gastric tube insertion between LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> and LMA Supreme<sup>TM</sup>.
- 3. To compare the laryngeal view of LMA Protector<sup>TM</sup>  $Cuff Pilot^{TM}$  and LMA Supreme<sup>TM</sup>.
- 4. To compare the complications in patients using LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> and LMA Supreme<sup>TM</sup>.

#### STUDY HYPOTHESIS

We hypothesised that LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> has similar OLP to LMA Supreme<sup>TM</sup>, is easily inserted with faster insertion time, and lesser complication.

#### **MATERIALS AND METHODS**

This prospective, single blinded, randomised controlled trial will be submitted for the approval of the Research Committee of Department of Anaesthesiology & Intensive Care, Universiti Kebangsaan Malaysia Medical Centre (UKMMC) and the Medical Research & Ethics Committee, UKMMC.

Patient information sheet (in Malay and English) will be given out and explained to patients. Written informed consent will be obtained from patients recruited into the study, which will be conducted by a single operator who has experience in insertion of both LMAs.

#### Study Site:

This proposed study will be carried out in operation theatres of Universiti Kebangsaan Malaysia Medical Centre.

## Inclusion Criteria:

- 1. Patients aged 18-65 years old.
- 2. Patients planned for general anaesthesia without muscle relaxant usage via SGA.

### **Exclusion Criteria:**

- 1. Patients with body mass index (BMI)  $> 35 \text{ kg/m}^2$ .
- 2. Patients with likelihood of difficult intubation (Simplified Airway Risk Index score  $\geq$  4). 13
- 3. Patients with increase risks of aspiration (gastro-oesophageal reflux disease, obstetric patients, hiatus hernia).

#### Methodology:

Patients who consented to the study will be randomized into 2 groups, Group P or Group S using an online Random Sequence Generator (https://www.random.org/sequences/). Patients in Group P will have LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> inserted during general anaesthesia whereas patients in Group S will receive LMA Supreme<sup>TM</sup>. The selection of SGA sizes will be done according to manufacturer's recommendation based on participant's weight. At the operating theatre, patients will be placed in supine position with a head rest. Standard monitoring consisting of pulse oximeter, non-invasive blood pressure (NIBP) and 3 lead electrocardiogram (ECG) will then be applied.

Both groups will receive similar induction regime which are: preoxygenation to achieve end-tidal fractional oxygen concentration > 0.85; intravenous (IV) fentanyl 1-2 mcg/kg; IV propofol 1.5-2.5 mg/kg and anaesthesia maintained with sevoflurane at minimum alveolar concentration (MAC) of 0.8-1.2 via manual mask ventilation with adjustable pressure limiting (APL) valve closed at < 20 cmH<sub>2</sub>O. Each SGA will be fully deflated and its posterior surface will be lubricated with water-based gel prior to placement. SGA will be inserted once participant's both pupils are in the centre and loss of motor response to jaw thrust. Both LMA Protector<sup>TM</sup> *Cuff Pilot*<sup>TM</sup> and LMA Supreme<sup>TM</sup> will be inserted using the single-handed rotational technique in the semi-sniffing position as recommended by manufacturer.

After insertion, the cuff in Group P will be insufflated with air till the cuff pilot valve is located in the centre of the green zone (estimated cuff pressure between 40-60 cmH<sub>2</sub>O). In Group S, the cuff will be insufflated with air in accordance to manufacturer's recommendation to 60 cmH<sub>2</sub>O by using a hand-held analog cuff pressure gauge (VBM *Medizintechnik GmbH*, Germany). The time to insertion - that is defined as duration from picking up the study device to presence of capnography tracing - will be recorded. The number of attempts will also be recorded. Any participant which require more than three attempts will be considered a fail attempt and will subsequently be managed appropriately by the attending anaesthetist.

After placement, a size 12-F gastric tube will be lubricated at the distal tip with water based lubricant and then inserted via the gastric channel of both groups. The number of attempt to insert a gastric tube will be recorded. Correct placement of the gastric tube will be determined by the detection of injected air through epigastric auscultation.

The position of SGA after insertion in relation to laryngeal inlet will be verified by passing an intubating bronchoscope to a position just proximal to the end of the SGA. The laryngeal view obtained at this point will be scored according to Keller *et al.*: Grade 1, clear view of the vocal cords; Grade 2, view of the arytenoids only; Grade 3, view of the epiglottis only; Grade 4, no laryngeal structures visible.<sup>14</sup>

Oropharyngeal leak pressure (OLP) will be assessed by setting the APL valve of the circle system at 40 cmH<sub>2</sub>O with fresh gas flow of 3 L/min. The OLP will be determined by observing the airway pressure at equilibrium until an audible noise is heard over the mouth with a stethoscope. For safety reasons, the maximum allowable OLP is 40 cmH<sub>2</sub>O.

Intraoperatively, anaesthesia will be maintained with sevoflurane at MAC of 0.8 to 1.2 in a mixture of 50% oxygen and 50% medical air with total flow of 2 L/min. Subsequent anaesthetic management including analgesia and anti-emetic will be in accordance to the discretion of the anaesthetist-in-charge.

SGA will be removed once patient awake and obeying simple commands. Presence of blood stain over the SGA will be recorded. Participants will be followed up in the recovery

and 6 hours after discharged from recovery to assess for presence of sore throat and hoarseness of voice.

#### STATISTICAL ANALYSIS

# Sample size calculation:

For the primary objective, we need 26 participants in each group to detect the difference of 4.5 cmH<sub>2</sub>O (20.7 vs 25.2 cmH<sub>2</sub>O) <sup>15</sup> with standard deviation of 5.7 at 80% power and alpha value of 0.05 using Power and Sample Size Calculation version 3.1.2.<sup>16</sup> With anticipation of 15% dropout rate, we decided to take a total of 60 participants.

# Statistical test:

All data will be entered into Microsoft Excel 2016 and analysed in Statistical Package for Social Science (SPSS) version 20.0. Result for the respective objectives will be analysed using the following statistical test and as appropriate. A value of p < 0.05 will be considered statistically significant.

| Results | Statistical analysis |
|------------------------------------------|------------------------|
| Assessing OLP | Student t-test |
| Comparing mean insertion time | Student <i>t</i> -test |
| Comparing ease of gastric tube insertion | Mann Whitney |
| Comparing laryngeal view | Mann Whitney |
| Comparing complications | Chi square |

#### **FLOW CHART**



# **GANTT CHART**

| Activity | Sep<br>17 | Oct -<br>Nov<br>17 | Dec 17 - May 18 | June -<br>Nov<br>18 | Dec<br>18 | Jan<br>19 | Feb -<br>Mar<br>19 | Apr<br>19 | May -<br>Jun 19 | Oct<br>19 |
|---|---|---|---|---|---|---|---|---|---|---|
| Proposal | | | | | | | | | | |
| presentation Quotation from LMA company Proposal editing and submission | | | | | | | | | | |
| Preparing research materials | | | | | | | | | | |
| Data collection | | | | | | | | | | |
| Data entry | | | | | | | | | | |
| Data analysis | | | | | | | *************************************** | | | |
| Study write up | | | | | | | | | | |
| Preliminary report | | | | | | | | | | |
| Final report presentation | | | | | | | | | | |
| Thesis submission | | | | | | | | | | |

# DATA COLLECTION SHEET

| Study No: | | Contact no: | | |
|---|---|---|---|---|
| 1. Demographic Data: | | | | |
| Name: | | | | |
| Age: | | Gender: Male / | Fema | ale |
| RN: | | ASA: I / II / | III | |
| Weight:kg | | Height: | cn | ı |
| Diagnosis: | | | | |
| Operation: | | | | |
| <ul> <li>2. Please circle the supraglottic LMA Supreme<sup>TM</sup> </li> <li>3. Duration of Insertion</li> </ul> | ` | GA) used: Protector <sup>TM</sup> Cuff P | ilot <sup>TM</sup> | |
| Time | Attempt No. 1 | Attempt No. 2 | Atte | mpt No. 3 |
| Duration (seconds) | | | - | |
| 4. Laryngeal view grade: 5. Oropharyngeal Leak Pressur | | cmH <sub>2</sub> O | | |
| 6. Gastric tube insertion attem | pt(s): | | | |
| 7. Total anaesthetic time (From | n induction to rem | oval of SGA): | | |
| 8. Postoperative Data | | | | |
| a) Presence of blood stain on | the SGA after rem | oval: Yes | / | No |
| b) Pharyngeal pain within 6 h | ours post op: | Yes | / | No |

#### REFERENCES

- 1. Van Zundert TCR V, Brimacombe JR, Ferson DZ, Bacon DR, Wilkinson DJ. Archie Brain: Celebrating 30 years of development in laryngeal mask airways. Anaesthesia. 2012;67(12):1375–85.
- 2. Brimacombe J. The advantages of the LMA over the tracheal tube or facemask: a meta-analysis. Can J Anaesth. 1995;42(11):1017–23.
- 3. Cook T, Howes B. Supraglottic airway devices: Recent advances. Contin Educ Anaesthesia, Crit Care Pain. 2011;11(2):56–61.
- 4. Miller DM. A proposed classification and scoring system for supraglottic sealing airways: A brief review. Anesth Analg. 2004;99(5):1553–9.
- 5. Teleflex. LMA Supreme<sup>TM</sup> A Second Generation SAD with and innovative Second Seal<sup>TM</sup> [Internet]. 2014 [cited 2017 Sep 19]. p. 1–2. Available from: http://www.teleflex.com/emea/documentLibrary/documents/940689-000001\_31817-LMA-TF-Supreme-A4\_1403\_PDF.pdf
- 6. Verghese C, Ramaswamy B. LMA-Supreme<sup>TM</sup> A new single-use LMA<sup>TM</sup> with gastric access: A report on its clinical efficacy. Br J Anaesth. 2008;101(3):405–10.
- 7. Teleflex. LMA Protector<sup>TM</sup> Instructions for use [Internet]. 2015 [cited 2017 Sep 19]. p. 1–16. Available from: http://www.lmaco-ifu.com/sites/default/files/node/1928/ifu/revision/3285/pbe2100000b-lma-protector-ifuuk.pdf
- 8. Bick E, Bailes I, Patel A, Brain AIJ. Fewer sore throats and a better seal: why routine manometry for laryngeal mask airways must become the standard of care. Anaesthesia [Internet]. 2014;69(12):1304–8. Available from: http://doi.org/10.1111/anae.12902
- 9. Asai T, Howell TK, Koga K, Morris S. Appropriate size and inflation of the laryngeal mask airway. Br J Anaesth. 1998;80(4):470–4.
- 10. Tiefenthaler W, Eschertzhuber S, Brimacombe J, Fricke E, Keller C, Kaufmann M. A randomised, non-crossover study of the GuardianCPV??? Laryngeal Mask versus the LMA Supreme??? in paralysed, anaesthetised female patients. Anaesthesia. 2013;68(6):600–4.
- 11. Saracoglu A, Dal D, Pehlivan G, Gögüs FY. The Professional Experience of Anaesthesiologists in Proper Inflation of Laryngeal Mask and Endotracheal Tube Cuff. Turkish J Anesth Reanim [Internet]. 2014;42(5):234–8. Available from: http://jtaics.org/jvi.aspx?pdir=tard&plng=eng&un=TARD-87487&look4=

- 12. Van Zundert AAJ, Skinner MW, Van Zundert TCR V, Luney SR, Pandit JJ. Value of knowing physical characteristics of the airway device before using it. Br J Anaesth. 2016;117(1):12–6.
- 13. El-Ganzouri AR, McCarthy RJ, Tuman KJ, Tanck EN, Ivankovich AD. Preoperative airway assessment: predictive value of a multivariate risk index. Anesth Analg. 1996;82(6):1197–204.
- 14. Keller C, Brimacombe J, Puhringer F. A fibreoptic scoring system to assess the position of laryngeal mask airway devices. Interobserver variability and a comparison between the standard, flexible and intubating laryngeal mask airways. Anasthesiol Intensivmed Notfallmedizin Schmerztherapie. 2000;35(11):692–4.
- 15. Zhang L, Seet E, Mehta V, Subramanyam R, Ankichetty SP, Wong DT, et al. Oropharyngeal leak pressure with the laryngeal mask airway Supreme at different intracuff pressures: a randomized controlled trial. Can J Anesth Can d'anesthésie [Internet]. 2011 Jul;58(7):624–9. Available from: https://doi.org/10.1007/s12630-011-9514-6
- 16. Dupont WD, Plummer WD. Power and sample size calculations for studies involving linear regression. Control Clin Trials. 1998;19(6):589–601.

# SIMPLIFIED AIRWAY RISK INDEX (SARI)

(El-Ganzouri et. al., 1996)

| Assessment | 0 point | 1 point | 2 points |
|---------------------------------|----------|--------------|----------|
| Interincisor gap | ≥ 4cm | < 4 cm | |
| Thyromental distance | > 6.5 cm | 6-6.5 cm | < 6 cm |
| Modified Mallampati Score | I-II | III | IV |
| Neck Movement | > 90 ° | 80-90 ° | < 80 ° |
| Ability to prognath | Yes | No | |
| Weight | < 90 kg | 90 - 110 kg | > 110 kg |
| History of difficult intubation | None | Questionable | Definite |

# Score:

< 4: unlikely to be difficult

 $\geq$  4: likely will be difficult